CLINICAL TRIAL: NCT01736813
Title: Treatment of Advanced Colorectal Cancer Patients With Hepatic Liver Metastases Using the CCR5-Antagonist Maraviroc (Phase I Maracon Trial)
Brief Title: CCR5-blockade in Metastatic Colorectal Cancer
Acronym: MARACON
Status: Completed | Type: Observational
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Other Study IDs: MARACON-001; 2012-000861-18 (EudraCT Number)
Record Dates: First submitted 2012-10-24; First posted 2012-11-29 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2014-07

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis; Liver Metastases
Keywords: colorectal cancer; liver metastases; chemotherapy; chemokine; CCR5 inhibition
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Maraviroc

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies, Serum and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CCR5-inhibitor at 300 mg/bid: colorectal cancer patients with liver metastases (twelve patients treated with 300 mg/bid)
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Twelve patients with 300 mg/bid
  Other Names: Celsentri

SUMMARY:
The surface molecule CCR5 is found on tumor cells within liver metastases of colorectal cancer. Inhibition of this molecule leads to a reduction in growth signals for tumor cells and subsequent slowed or halted tumor growth. The agent for the inhibition of CCR5 has already received FDA approval for treatment of HIV and has shown little side effects and toxicities even on long term treatment. Therefore CCR5-inhibition has the potential of providing non-toxic tumor growth inhibition.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent (must be available before enrollment in the trial)
* age ≥ 18 years
* male or female patient with a history of treated metastatic stage IV colorectal cancer with liver metastases of the primary colorectal cancer
* histologically confirmed liver metastasis of colorectal cancer with histologically confirmed CCR5 (C-C chemokine receptor type 5) expression in the tumor cells
* expected survival of at least three months
* Karnofsky performance status > 70 %
* patients that have received current standard treatment options (progression or intolerance to oxaliplatin, irinotecan and 5-Fluorouracil with or without treatment combinations of cetuximab and/or bevacizumab or panitumumab)
* no chemotherapy treatment within the last three weeks
* within the last 2 weeks prior to study day 1 the following laboratory parameters, which should be within the ranges specified (or as deemed acceptable by trial investigator): absolute neutrophil count (ANC) ≥ 1000/mm3 (≥ 1.0 x 109/L), platelets ≥ 80.000/mm3 (≥ 80 x 109/L), creatinine Clearance limit as assessed by glomerular filtration rate > 60 mL/min/1.73m², ALT (alanine transaminase), AST (aspartate transaminase), and total bilirubin all ≤ 5.0 x ULN (upper limit normal)
* able and willing to give valid written informed consent and to understand character and individual consequences of the clinical trial
* if the patient is female, she must be of non-childbearing potential, or practice adequate contraception.

Exclusion Criteria:

* Patients with severe kidney disorders (GFR of <30 mL/min/1.73m² and diagnosed kidney disease) or who are on hemodialysis. The patient requires concomitant chronic treatment with systemic corticosteroids or any other immunosuppressive agents. Topical or inhalational steroids are permitted.
* Patients taking immunomodulatory medication (Type 1 interferons).
* Use of any investigational or non-registered product (drug or vaccine) other than the study treatment
* Patients with single metastatic lesions (intent to resect the metastasis)
* Patients with metastatic colorectal cancer that have a drastic clinical progression (e.g. from Karnofsky performance 100% to 60%) within the last six weeks before screening cannot participate
* The patient has a history of autoimmune disease.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other chronic infections (HBV, HCV).or has another confirmed or suspected immunosuppressive or immunodeficient condition.
* The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
* The patient has concurrent chronic severe medical problems (heart failure, uncontrolled diabetes, bleeding disorder etc.), unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* The patient has previous or concomitant malignancies at other sites, except effectively treated carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* For female patients: the patient is pregnant or lactating.
* Women of childbearing potential: Refusal or inability to use effective means of contraception
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Participation in other clinical trials or observation period of competing trials, respectively
* No subject will be allowed to enroll in this trial more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: large university hospital with local private practice referrers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
safety as occurence of adverse events ≥ Grade 3 according to CTCAE, Version 4.0 criteria, that are definitely, probably, or possible related to the administration of the investigational agent | after eight weeks of treatment
  safety, tolerability and feasibility will be assessed after eight weeks of continuous intake of the CCR5-inhibitor. Safety measures include blood analyses (hematologic, liver function, renal function etc.) and the overall performance status of the patient. Especially infections and infection-related events are investigated.

SECONDARY OUTCOMES:
Progression Free Survival | one year after eight weeks of treatment
  Patients will be evaluated for one year afterwards to assess progression free survival.
Tumor response according to the Response Evaluation Criteria in Solid Tumors (RECIST) | after eight weeks of treatment
  Tumor response will be evaluated after eight weeks of continuous treatment with the CCR5-inhibitor, using the RECIST criteria on MRI images (comparing pre- and post-treatment)
Tissue level responses of growth inhibition via the CCR5 axis | during the first four weeks of treatment
  The evaluation of tissue alterations within the tumor microenvironment induced by CCR5-inhibition will be performed during the first four weeks of treatment, comparing the pre-treatment tissue situation with the post-treatment situation.
Overall survival | one year after eight weeks of treatment
  Patients will be evaluated for one year afterwards to assess overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Halama, MD, Principal Investigator — National Center for Tumor Diseases (NCT), University Hospital Heidelberg, Heidelberg, Germany; Dirk Jaeger, MD, Study Director — National Center for Tumor Diseases (NCT), University Hospital Heidelberg, Germany
Locations (1):
- National Center for Tumor Diseases, Department of Medical Oncology, Heidelberg, Baden-Wurttemberg, Germany

REFERENCES:
- [Result] Halama N, Zoernig I, Berthel A, Kahlert C, Klupp F, Suarez-Carmona M, Suetterlin T, Brand K, Krauss J, Lasitschka F, Lerchl T, Luckner-Minden C, Ulrich A, Koch M, Weitz J, Schneider M, Buechler MW, Zitvogel L, Herrmann T, Benner A, Kunz C, Luecke S, Springfeld C, Grabe N, Falk CS, Jaeger D. Tumoral Immune Cell Exploitation in Colorectal Cancer Metastases Can Be Targeted Effectively by Anti-CCR5 Therapy in Cancer Patients. Cancer Cell. 2016 Apr 11;29(4):587-601. doi: 10.1016/j.ccell.2016.03.005. PMID 27070705